CLINICAL TRIAL: NCT00450736
Title: A Phase I Trial of Postoperative Radiation With Dose-Escalation of A Cox-2 Inhibitor, Celebrex™ (CELECOXIB) in Patients With Soft Tissue Sarcoma of the Extremity
Brief Title: Celecoxib and Radiation Therapy in Treating Patients With Stage II or Stage III Soft Tissue Sarcoma of the Arm, Hand, Leg, or Foot That Has Been Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030283; SCCC-2003053 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20051240 (Other: Western Institution Reviw Board)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Childhood Malignant Fibrous Histiocytoma of Bone; Sarcoma
Keywords: chondrosarcoma; adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; childhood angiosarcoma; childhood fibrosarcoma; childhood leiomyosarcoma; childhood liposarcoma; childhood neurofibrosarcoma; childhood synovial sarcoma; nonmetastatic childhood soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; childhood malignant hemangiopericytoma; localized childhood malignant fibrous histiocytoma of bone
MeSH Terms: conditions — Sarcoma; Chondrosarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant | interventions — Celecoxib; Chemotherapy, Adjuvant; Radiotherapy

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: celecoxib; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: celecoxib
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving celecoxib together with radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I trial is studying the side effects and best dose of celecoxib when given together with radiation therapy in treating patients with stage II or stage III soft tissue sarcoma of the arm, hand, leg, or foot that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of adjuvant celecoxib administered with radiotherapy in patients with resected stage II or III soft tissue sarcoma of the extremity.

OUTLINE: This is a dose-escalation study of celecoxib.

Beginning within 10 weeks of the most recent resection, patients undergo standard radiotherapy once daily, 5 days a week, in weeks 1-7. Patients also receive oral celecoxib twice daily in weeks 1-7 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of celecoxib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. A maximum of 6 patients are treated at the MTD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma of the extremity, including the following disease types:

  * Liposarcoma
  * Leiomyosarcoma
  * Synovial cell sarcoma
  * Malignant fibrous histiocytoma
  * Spindle cell sarcoma
  * Fibrosarcoma
  * Chondrosarcoma
  * Angiosarcoma
  * Hemangiopericytoma
  * Neurofibrosarcoma
* The following disease types are excluded:

  * Kaposi's sarcoma
  * Rhabdomyosarcoma
  * Dermatofibrosarcoma
  * Epithelioid cell sarcoma
  * Ewing's sarcoma
  * Osteosarcoma
* Intermediate- or high-grade tumor ≥ 5.0 cm in 1 dimension (stage II or III disease)
* Locally resected disease

  * One prior wide local excision of the sarcoma in the same location of the extremity within the past 6 months allowed
  * Prior neoadjuvant chemotherapy (of ≤ 3 courses), followed by a limb-sparing surgical resection of sarcoma found to have < 90% pathological tumor necrosis allowed
  * Prior resection of an extremity mass that is subsequently found to be a sarcoma meeting study criteria, followed by ≤ 3 courses of chemotherapy (independent of the percentage of pathological tumor necrosis) allowed
* No evidence of nodal or distant metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* WBC ≥ 3,000/mm³
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* SGPT and SGOT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Calcium ≤ 1.3 times ULN
* No prior malignancy except cutaneous nonmelanomatous skin cancer, carcinoma in situ of the cervix, or other cancer for which the patient has been disease-free for at least 5 years
* No history of allergic reaction to sulfonamides or NSAIDs
* No known hypersensitivity to celecoxib or any component of its formulation
* No known HIV positivity
* No known coronary artery disease
* No cardiac event of any kind within the past 6 months
* No concurrent unstable cardiac status
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the extremity requiring radiation for this study
* No prior systemic chemotherapy for a malignant tumor
* No concurrent dilantin or lithium carbonate
* No other concurrent prescription or over-the-counter nonsteroidal anti-inflammatory agents (NSAIDs)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Local failure | 3 years
Regional relapse | 3 years
Distant failure | 3 years
Overall survival | 3 years
Progression-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aaron H. Wolfson, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States